CLINICAL TRIAL: NCT03261635
Title: Prospective Randomized Controlled Trial of Combination Ranibizumab and Indomethacin for Exudative Age-Related Macular Degeneration
Brief Title: Ranibizumab Plus Indomethacin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Andrea Russo, Principal Investigator, Università degli Studi di Brescia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSAIDs_02
Record Dates: First submitted 2017-08-20; First posted 2017-08-25 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Macular Edema
MeSH Terms: conditions — Macular Edema | interventions — Ranibizumab; Indomethacin

STUDY DESIGN:
Intervention Model Description: This was a prospective, randomized, pilot study in 58 patients with naï ve CNV. Patients were randomized 1:1 into 2 groups: ranibizumab monotherapy (RM group) and ranibizumab plus indomethacin (RI group). All patients received monthly 0.5 mg ranibizumab intravitreal injections for 3 months, after which monthly injections were administered pro re nata. RI patients also self- administered one drop of indomethacin three times a day for 12 months. All patients were followed up for 12 months.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ranibizumab Monotherapy (Active Comparator): All patients received monthly 0.5 mg ranibizumab intravitreal injections for 3 months, after which monthly injections were administered pro re nata
  Interventions: Drug: Ranibizumab Injection
- Ranibizumab + Indomethacin (Experimental): All patients received monthly 0.5 mg ranibizumab intravitreal injections for 3 months, after which monthly injections were administered pro re nata. Moreover, patients also self- administered one drop of indomethacin three times a day for 12 months. All patients were followed up for 12 months.
  Interventions: Drug: Ranibizumab Injection; Drug: Indomethacin

INTERVENTIONS:
Drug: Ranibizumab Injection — patients received monthly 0.5 mg ranibizumab intravitreal injections for 3 months, after which monthly injections were administered pro re nata
Drug: Indomethacin — patients self-administered one drop of indomethacin 0.5% eye drops three times a day for 12 months
  Arms: Ranibizumab + Indomethacin

SUMMARY:
To evaluate whether indomethacin eyedrops plus intravitreal ranibizumab (IVR) provides additional benefit over IVR monotherapy for treatment of choroidal neovascularization (CNV) in age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* provision of written informed consent and compliance with study assessments for the full duration of the study
* age > 40 years
* presence of treatment-naïve neovascular AMD.

Exclusion Criteria:

* any previous intravitreal treatment
* previous laser treatment in the study eye
* myopia > 7 diopters in the study eye
* concurrent eye disease in the study eye that could compromise visual acuity (e.g., diabetic retinopathy and advanced glaucoma)
* concurrent corneal epithelial disruption or any condition that would affect the ability of the cornea to heal
* known sensitivity to any component of the formulations being investigated.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-01-07 (Actual); Primary Completion 2016-12-07 (Actual); Study Completion 2017-07-25 (Actual)

PRIMARY OUTCOMES:
Central Retinal Thickness (microns) | 12-month
  Optical Coherence Tomography will be used to assess central retinal thickness.
Visual Acuity (LogMAR) | 12-month
  ETDRS charts will be used to assess best corrected visual acuity

IPD SHARING:
Plan to Share IPD: No